CLINICAL TRIAL: NCT04941963
Title: Functional Evaluation of the Diaphragm With Bedside Ultrasound in Infants With Bronchopulmonary Dysplasia: a Single Centre Prospective Trial
Brief Title: Ultrasound Assessment of Diaphragmatic Function in Infants With BPD
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0224-E
Record Dates: First submitted 2021-05-20; First posted 2021-06-28 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2021-10

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: preterm; neonates; Mechanical ventilation; Bronchopulmonary Dysplasia; Chest; Ultrasound
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Chest ultrasound — Patients will undergo chest ultrasound scanning after obtaining parent's consent. each enrolled patient will have one chest ultrasound to assess diaphragmatic function and lung ultrasound severity score.

SUMMARY:
Preterm infants have high and prolonged exposure to positive pressure ventilation, which contributes to acute lung injury and the development of bronchopulmonary dysplasia (BPD). Despite the risk of diaphragmatic dysfunction in infants with BPD, the effect of prolonged ventilator support on the diaphragmatic function of preterm infants has not been well characterized.

Hence, we aim to characterize the diaphragmatic function of very preterm neonates with BPD who are corrected to ≥ 36 weeks using bedside ultrasound in comparison to healthy newborns born at ≥ 36 weeks gestation.

DETAILED DESCRIPTION:
Study Design and setting; This is a prospective descriptive pilot study that will be conducted on infants born at ≤ 32 weeks gestation who meet eligibility criteria and are admitted to the neonatal intensive care at Mount Sinai Hospital and healthy newborns born at at ≥ 36 weeks gestation. Enrollment of eligible infants will start after obtaining approval from the Research Ethics Board at Mount Sinai Hospital and parental consent.

Time of assessment; Parents of infants who are eligible for the study will be approached for consent. Chest ultrasound (lung ultrasound and diaphragmatic function assessment) will be performed at ≥ 36 weeks corrected gestational age. Chest ultrasound will be done before a feeding to avoid any concerns of a full stomach on diaphragmatic assessment.

Study procedure; Functional assessment of the diaphragm will be done by two of the investigators. Standard variables for assessing diaphragm function will be used including diaphragmatic thickness, diaphragmatic thickness fraction, and diaphragmatic excursion (DE). Diaphragmatic thickness fraction, and diaphragmatic excursion will be calculated. Inter-rater agreement will be assessed using raw percentage of agreement (Pa), Cohen's and Kappa (κ), and G wet agreement coefficient (AC1). Intra-class correlation (ICC) will be determined for variables with continuous measurements (mixed factorial design). High-resolution linear and curvilinear US probes of 20-5 and 10-3 MegahertZ will be used to measure diaphragmatic thickness fraction, and diaphragmatic excursion [amplitude] respectively using both B and M modes.

Diaphragmatic assessment technique; Diaphragm assessment will be performed in the supine position. To measure diaphragmatic excursion, the curvilinear probe will be placed on the lower intercostal spaces between the mid-clavicular and anterior axillary lines on the right side. Using the B mode, the proper exploration line of the diaphragm will be detected by directing the beam perpendicular to the posterior third of the right hemidiaphragm. By M mode, the cyclic caudal diaphragmatic displacement with respiration will be measured as the perpendicular distance between the most caudal point of the liver or spleen at the end of expiration and the end of inspiration. The average of three respiratory cycles will be taken.

The assessment of the diaphragmatic efficiency as a pressure generator will be evaluated using the diaphragmatic thickness fraction. Diaphragmatic thickness will be measured at the apposition zone which can be obtained by placing the linear transducer above the 10th rib in the mid-axillary or anterior axillary lines in the right intercostal spaces. By B mode, three distinct layers will be seen, the diaphragm as a hypo-echoic area bordered by two clear echogenic lines of the pleural membrane (upper line) and the peritoneal membrane (lower line). Using M-mode tracing, inspiratory diaphragmatic thickness will be measured as the maximum perpendicular distance between pleural and peritoneal layers and by the same way expiratory diaphragmatic thickness will be recorded. diaphragmatic thickness fraction will be calculated using the following formula:

diaphragmatic thickness fraction = [(inspiratory thickness - expiratory thickness)/expiratory thickness] x 100.

The average of the calculated diaphragmatic thickness fraction from three respiratory cycles will be estimated. The higher scores the better the diaphragmatic function. All Chest ultrasound assessments will be undertaken using a standard aseptic technique.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Infants who are born at ≤ 32 weeks gestation,
* Admitted to the neonatal intensive care at Mount Sinai Hospital
* Receiving oxygen or respiratory support at ≥ 36 weeks gestation

Control:

* Infants who are born at ≥ 36 weeks gestation
* Admitted to the level 1 nursery.
* Informed consent obtained from parents or guardians prior to enrolment in the study.

Exclusion Criteria:

* Infants who have congenital or chromosomal abnormalities.
* Parents declined the consent.

Min Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants who are born at ≤ 32 weeks gestation, admitted to the neonatal intensive care at Mount Sinai Hospital, and receiving oxygen or respiratory support at ≥ 36 weeks gestation will be eligible for the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the diaphragmatic Thickness fraction and diaphragmatic excursion in neonates with bronchopulmonary dysplasia | 1 year
  * Chest ultrasound will be used to evaluate the diaphragmatic function in neonates at ≥ 36 weeks gestation with bronchopulmonary dysplasia in comparison to diaphragmatic function in healthy newborns born at ≥ 36 weeks gestation.
  * Assessment of Diaphragmatic Thickness in millimetres.
  * Assessment of Diaphragmatic Excursion in millimetres.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung T, Mohsen N, Ghanem M, Ibrahim J, Shah J, Kajal D, Shah PS, Mohamed A. Diaphragmatic Thickness and Excursion in Preterm Infants With Bronchopulmonary Dysplasia Compared With Term or Near Term Infants: A Prospective Observational Study. Chest. 2023 Feb;163(2):324-331. doi: 10.1016/j.chest.2022.08.003. Epub 2022 Aug 10. PMID 35963296